CLINICAL TRIAL: NCT06847230
Title: How Does DT1 Sphere Perform in Current and Successful Acuvue MAX Wearers?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07-01CL
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Contact Lens Comfort and Successful Refitting
Keywords: Contact lenses; Contact lens comfort

STUDY DESIGN:
Intervention Model Description: This 2-week, 3-visit clinical study will refit current Acuvue Max contact lens wearers into Dailies Total 1 contact lenses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dailies total 1 contact lenses (Experimental): Acuvue max wearers will be refit into dailies total 1
  Interventions: Device: Dailies total 1 contact lenses

INTERVENTIONS:
Device: Dailies total 1 contact lenses — successful refit into dt1 will be determined

SUMMARY:
The goal of this prospective study is to to understand if satisfied MAX Contact lens (CL)wearers can be successfully refit into Dailies total 1 (DT1) CL in healthy MAX CL wearers between the ages of 18-40. The main question is to determine the number of participants who can successfully be re-fit into DT1 CL, by utilizing a cldeq-8 questionnaire as well as an investigator developed questionnaire to gauge comfort and satisfaction.

ELIGIBILITY:
* Inclusion Criteria:
* Adults, 18- to 40-year-old, Oasys MAX 1-day CL wearers with best-corrected 20/20 visual acuity or better.
* Participants will be required to have worn Oasys MAX 1-day CLs for at least 3 months in the past year and currently wearing these CLs.
* All participants will be required to have a CLDEQ-8 score <12 while wearing their habitual CLs (Oasys MAX 1-days) and to indicate that they are satisfied with Oasys MAX 1-day CLs (Yes/No).
* Participants will be required to be able to wear DT1 Sphere CLs (astigmatism < 0.75D OD/OS).
* Participants will be required to wear the study CLs for ≥12 hours with no overnight wear
* Participants will be required to use digital devices at least 8 hours/day.
* Participants will be required to provide a glasses prescription that is less than 3 years old.
* Exclusion Criteria:
* Have presbyopia and/or need a reading add as determined during their initial manifest refraction.
* Have worn DT1 in the past for more than 1 week.
* Are past rigid CL wearers.
* Have a history of being diagnosed with dry eye or ocular allergies.
* Have known systemic health conditions that are thought to alter tear film physiology.
* Have corrected acuity 1 line or more worse vision recorded at Visit 2 (compared to the Visit 1 findings) with their optimized Oasys MAX 1-day lenses.
* Have a history of viral eye disease.
* Have a history of ocular surgery.
* Have a history of severe ocular trauma.
* Have a history of corneal dystrophies or degenerations.
* Have active ocular infection or inflammation.
* Are currently using isotretinoin-derivatives or ocular medications.
* Are pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Likelihood of continuing to wear DT1 | 3 weeks
  A Likert questionnaire will be used to determine patient-reported outcomes -50 being uncomfortable and 50 being extremely comfortbale
Overall satisfaction while wearing DT1 | 3 weeks
  A Likert questionnaire will be used to determine patient-reported outcomes. With answers that are positive such as strongly agree to product satisfaction are better.

CONTACTS AND LOCATIONS:
Locations (1):
- The Southern College of Optometry, Memphis, Tennessee, United States